CLINICAL TRIAL: NCT02949154
Title: Elevated LDH Serum Levels and FDG-PET in Metastatic Melanoma Patients
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201600693
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metastatic melanoma patients: All patients >18 years with histologically proven metastatic melanoma (American Joint Committee on Cancer [AJCC] stage IV melanoma) treated in the UMCG between May 2014 and December 2015.

SUMMARY:
A retrospective study investigating the relationship between FDG-PET uptake and LDH levels.

DETAILED DESCRIPTION:
Patient characteristics, tumour characteristics including the BRAF mutation status and baseline serum S100B and LDH levels of each patient will be retrospectively determined from the electronical patient file. In each patient, tumour burden and 18F-FDG uptake of the tumour lesions will be measured using multiple standard quantification parameters of the baseline 18F-FDG-PET scan. Tumour burden will also be measured on the baseline contrast enhanced CT scan. The correlation of each FDG-PET parameter with baseline LDH and S100B levels, respectively, will be analyzed using univariate and multivariate regression analysis.

ELIGIBILITY:
Inclusion Criteria:

- All patients >18 years with histologically proven metastatic melanoma (American Joint Committee on Cancer [AJCC] stage IV melanoma) treated in the UMCG between May 2014 and December 2015.

Exclusion Criteria:

* participation in interventional studies
* missing baseline 18F-FDG PET scan and/or baseline contrast enhanced CT scan
* missing baseline serum LDH level
* missing BRAF mutation status, concurrent malignancies or a history of previous malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic melanoma
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Independent correlation between baseline serum LDH level and 18F-FDG uptake of tumour lesions | 3 months

SECONDARY OUTCOMES:
Correlation between baseline serum LDH level and tumour 18F-FDG uptake in subgroups separated by metastasis site | 3 months
Correlation between baseline serum S100B level and tumour 18F-FDG uptake | 3 months
Difference between tumour burden as measured on CT scan and on 18F-FDG-PET | 3 months
Difference between tumour volume as determined by manual measurement or semiautomatic measurement | 3 months
Correlation of baseline serum LDH level with tumour volume as measured on CT scan and as measured on 18F-FDG-PET scan | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Jalving, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No